CLINICAL TRIAL: NCT03954834
Title: A Randomized, Double-blind, Placebo-Controlled Trial Comparing the Efficacy and Safety of Three Tirzepatide Doses Versus Placebo in Patients With Type 2 Diabetes, Inadequately Controlled With Diet and Exercise Alone
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes Not Controlled With Diet and Exercise Alone
Acronym: SURPASS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17000; I8F-MC-GPGK (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: glucose-dependent insulinotropic polypeptide (GIP); glucagon-like peptide-1 (GLP-1); GIP/GLP-1 dual receptor agonist; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Tirzepatide (Experimental): Participants received 5 milligrams (mg) of tirzepatide as subcutaneous injection once a week.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): Participants received 10mg of tirzepatide as subcutaneous injection once a week.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): Participants received 15mg of tirzepatide as subcutaneous injection once a week.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received placebo as subcutaneous injection once a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The goal for this study is to evaluate the efficacy and safety of tirzepatide versus placebo in participants with type 2 diabetes not under control with diet and exercise alone. The study will last approximately 47 weeks and may include about 15 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus (T2DM).
* Are naïve to diabetes injectable therapies and have not used any oral antihyperglycemic medications (OAMs) during the 3 months preceding screening.
* Have HbA1c between ≥7.0% and ≤9.5%.
* Be of stable weight (± 5%) for at least 3 months before screening.
* Have a BMI ≥23 kilograms per meter squared (kg/m²) at screening.

Exclusion Criteria:

* Have type 1 diabetes mellitus.
* Have had chronic or acute pancreatitis any time prior to study entry.
* Have proliferative diabetic retinopathy or diabetic maculopathy or nonproliferative diabetic retinopathy requiring acute treatment.
* Have disorders associated with slowed emptying of the stomach, or have had any stomach surgeries for the purpose of weight loss.
* Have an estimated glomerular filtration rate <30 mL/minute/1.73 m².
* Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months.
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2.
* Have been taking weight loss drugs, including over-the-counter medications during the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (53):
- United States (28):
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Valley Clinical Trials, Inc., Northridge, California
  - National Research Institute, Panorama City, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Encore Medical Research, LLC, Hollywood, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - South Florida Wellness & Clinical Research Institute, Margate, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Agile Clinical Research Trials, Atlanta, Georgia
  - Sky Clinical Research Network, Atlanta, Georgia
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Clinical Research Professionals, Chesterfield, Missouri
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Aventiv Research, Columbus, Ohio
  - Intend Research, Norman, Oklahoma
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Capital Clinical Research Center, Olympia, Washington
  - Rockwood Clinic Research Center, Spokane, Washington
- India (9):
  - Dr. Jivraj Mehta Smarak Health Foundation, Ahmedabad, Gujarat
  - Bangalore Medical College and Research Institute, Bangalore, Karnataka
  - M S Ramaiah Medical College Hospital, Bangalore, Karnataka
  - BSES Municipal General Hsptl, Mumbai, Maharashtra
  - Ruby Hall Clinic and Grant Medical Foundation, Pune, Maharashtra
  - Vijay Vallabh Hospital, Virār, Maharashtra
  - Lifepoint Multispecialty Hsptl, Wakad, Pune
  - Ramdevrao Hospital, Hyderabad, Telangana
  - Gandhi Hospital, Telangana
- Japan (10):
  - Minamiakatsuka Clinic, Mito, Ibaraki
  - Takai Naika Clinic, Kamakura, Kanagawa
  - Tsuruma Kaneshiro Diabetes Clinic, Yamato, Kanagawa
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Meiwa Hospital, Chiyodaku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Tokyo Center Clinic, Chuo-ku, Tokyo
  - IHL Shinagawa East One Medical Clinic, Minato-ku, Tokyo
  - Sato Naika Clinic, Ōta-ku, Tokyo
- Mexico (4):
  - Hospital Universitario UANL, Monterrey, Nuevo León
  - Unidad Medica para la Salud Integral (UMSI), Monterrey, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasc, Madero, Tamaulipas
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
- Puerto Rico (2):
  - GCM Medical Group PSC, San Juan, PR
  - Clinical Research Puerto Rico, Inc., San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] De Block C, Peleshok J, Wilding JPH, Kwan AYM, Rasouli N, Maldonado JM, Wysham C, Liu M, Aleppo G, Benneyworth BD. Post Hoc Analysis of SURPASS-1 to -5: Efficacy and Safety of Tirzepatide in Adults with Type 2 Diabetes are Independent of Baseline Characteristics. Diabetes Ther. 2025 Jan;16(1):43-71. doi: 10.1007/s13300-024-01660-0. Epub 2024 Nov 12. PMID 39531161
- [Derived] Boye KS, Sapin H, Dong W, Williamson S, Lee CJ, Thieu VT. Improved Glycaemic and Weight Management Are Associated with Better Quality of Life in People with Type 2 Diabetes Treated with Tirzepatide. Diabetes Ther. 2023 Nov;14(11):1867-1887. doi: 10.1007/s13300-023-01457-7. Epub 2023 Sep 5. PMID 37668888
- [Derived] Boye KS, Thieu VT, Sapin H, Lee CJ, Lando LF, Brown K, Bray R, Wiese RJ, Patel H, Rodriguez A, Yu M. Patient-Reported Outcomes in People with Type 2 Diabetes Receiving Tirzepatide in the SURPASS Clinical Trial Programme. Diabetes Ther. 2023 Nov;14(11):1833-1852. doi: 10.1007/s13300-023-01451-z. Epub 2023 Aug 1. PMID 37526908
- [Derived] Sattar N, McGuire DK, Pavo I, Weerakkody GJ, Nishiyama H, Wiese RJ, Zoungas S. Tirzepatide cardiovascular event risk assessment: a pre-specified meta-analysis. Nat Med. 2022 Mar;28(3):591-598. doi: 10.1038/s41591-022-01707-4. Epub 2022 Feb 24. PMID 35210595
- [Derived] Rosenstock J, Wysham C, Frias JP, Kaneko S, Lee CJ, Fernandez Lando L, Mao H, Cui X, Karanikas CA, Thieu VT. Efficacy and safety of a novel dual GIP and GLP-1 receptor agonist tirzepatide in patients with type 2 diabetes (SURPASS-1): a double-blind, randomised, phase 3 trial. Lancet. 2021 Jul 10;398(10295):143-155. doi: 10.1016/S0140-6736(21)01324-6. Epub 2021 Jun 27. PMID 34186022
- See also: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes Not Controlled With Diet and Exercise Alone (SURPASS-1) — https://www.lillytrialguide.com/en-US/studies/adult-type-2-diabetes/GPGK#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mg Tirzepatide: Participants received 5 mg of tirzepatide as subcutaneous injection once a week.
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Started | 121 | 121 | 121 | 115
Received at Least One Dose of Study Drug | 121 | 121 | 121 | 115
Completed | 114 | 112 | 103 | 99
Not Completed | 7 | 9 | 18 | 16
Not completed — Adverse Event | 1 | 3 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 13 | 6
Not completed — Participant left the country | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 2 | 3 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 121 | 121 | 121 | 115 | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.10 (11.88) | 55.80 (10.35) | 52.90 (12.34) | 53.60 (12.79) | 54.10 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 49 | 58 | 59 | 231
  Male | 56 | 72 | 63 | 56 | 247
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 54 | 55 | 48 | 207
  Not Hispanic or Latino | 48 | 49 | 42 | 45 | 184
  Unknown or Not Reported | 23 | 18 | 24 | 22 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 31 | 31 | 30 | 26 | 118
  Asian | 45 | 43 | 42 | 38 | 168
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 6 | 5 | 22
  White | 38 | 43 | 43 | 46 | 170
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 18 | 20 | 18 | 17 | 73
  Japan | 23 | 22 | 23 | 21 | 89
  Mexico | 42 | 40 | 42 | 40 | 164
  Puerto Rico | 2 | 4 | 5 | 1 | 12
  United States | 36 | 35 | 33 | 36 | 140
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.97 (0.841) | 7.90 (0.78) | 7.85 (1.02) | 8.05 (0.80) | 7.94 (0.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Prior Use of oral antihyperglycemic medication (OAM) (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline value, excluding patients discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 121 | 118 | 116 | 112
Percentage of HbA1c | -1.87 (0.094) | -1.89 (0.096) | -2.07 (0.098) | 0.04 (0.105)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.91, 95% CI 2-sided [-2.18 to -1.63]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.93, 95% CI 2-sided [-2.21 to -1.65]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -2.11, 95% CI 2-sided [-2.39 to -1.83]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Prior Use of OAM (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 121 | 118 | 116 | 112
Kilograms (kg) | -7.0 (0.52) | -7.8 (0.53) | -9.5 (0.54) | -0.7 (0.57)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.3, 95% CI 2-sided [-7.8 to -4.7]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.1, 95% CI 2-sided [-8.6 to -5.5]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -8.8, 95% CI 2-sided [-10.3 to -7.2]

3. Secondary Outcome: Percentage of Participants With HbA1c Target Value of <7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 121 | 118 | 116 | 112
Percentage of participants | 86.78 | 91.53 | 87.93 | 19.64
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 49.00, 95% CI 2-sided [21.12 to 113.67]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 80.39, 95% CI 2-sided [31.80 to 203.19]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 52.95, 95% CI 2-sided [22.30 to 125.73]

4. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: Fasting serum glucose (FSG) is a test to determine sugar levels in serum sample after an overnight fast. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Prior Use of OAM (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per Deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 121 | 118 | 116 | 112
milligram per Deciliter (mg/dL) | -43.6 (3.40) | -45.9 (3.45) | -49.3 (3.62) | 12.9 (4.00)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.776, Mixed Models Analysis; LS Mean Difference = -1.5, 95% CI 2-sided [-11.9 to 8.9]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.622, Mixed Models Analysis; LS Mean Difference = -2.6, 95% CI 2-sided [-13.0 to 7.8]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.908, Mixed Models Analysis; LS Mean Difference = -0.6, 95% CI 2-sided [-11.1 to 9.8]

5. Secondary Outcome: Percentage of Participants With HbA1c Target Value of <5.7%
Description: as for outcome 3
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 121 | 118 | 116 | 112
Percentage of participants | 33.88 | 30.51 | 51.72 | 0.89
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 40.28, 95% CI 2-sided [7.74 to 209.71]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 34.12, 95% CI 2-sided [6.53 to 178.19]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 85.13, 95% CI 2-sided [16.36 to 443.13]

6. Secondary Outcome: Mean Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Postmeal, Midday Premeal, Midday 2-hour Postmeal, Evening Premeal, Evening 2-hour Postmeal and Bedtime. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Prior Use of OAM (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 115 | 111 | 108 | 101
mg/dL
  Morning Premeal - Fasting | -46.9 (2.09) | -47.9 (2.11) | -45.7 (2.23) | -9.2 (2.53)
  Morning 2-hour Postmeal: number analyzed (Participants) | 115 | 111 | 107 | 101
  Morning 2-hour Postmeal | -69.5 (3.41) | -61.4 (3.44) | -68.9 (3.66) | -11.6 (4.12)
  Midday Premeal | -43.5 (2.80) | -42.5 (2.82) | -42.7 (3.00) | -2.6 (3.42)
  Midday 2-hour Postmeal | -64.2 (3.60) | -60.0 (3.63) | -63.4 (3.84) | -12.7 (4.33)
  Evening Premeal: number analyzed (Participants) | 115 | 111 | 106 | 101
  Evening Premeal | -44.8 (2.80) | -45.1 (2.82) | -42.3 (3.02) | -5.8 (3.38)
  Evening 2-hour Postmeal: number analyzed (Participants) | 115 | 110 | 107 | 100
  Evening 2-hour Postmeal | -61.9 (3.76) | -62.8 (3.81) | -63.5 (4.03) | -10.3 (4.52)
  Bedtime: number analyzed (Participants) | 113 | 108 | 108 | 101
  Bedtime | -57.0 (3.49) | -59.8 (3.52) | -60.8 (3.66) | -9.1 (4.10)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Morning Premeal - Fasting; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -37.7, 95% CI 2-sided [-44.1 to -31.2]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Morning Premeal - Fasting; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -38.6, 95% CI 2-sided [-45.1 to -32.2]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Morning Premeal - Fasting; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -36.5, 95% CI 2-sided [-43.1 to -29.8]
Statistical Analysis 4: Comparison: 5 mg Tirzepatide vs Placebo; Morning 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -57.9, 95% CI 2-sided [-68.4 to -47.4]
Statistical Analysis 5: Comparison: 10 mg Tirzepatide vs Placebo; Morning 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -49.7, 95% CI 2-sided [-60.3 to -39.2]
Statistical Analysis 6: Comparison: 15 mg Tirzepatide vs Placebo; Morning 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -57.3, 95% CI 2-sided [-68.1 to -46.4]
Statistical Analysis 7: Comparison: 5 mg Tirzepatide vs Placebo; Midday Premeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -40.9, 95% CI 2-sided [-49.6 to -32.2]
Statistical Analysis 8: Comparison: 10 mg Tirzepatide vs Placebo; Midday Premeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -39.9, 95% CI 2-sided [-48.6 to -31.2]
Statistical Analysis 9: Comparison: 15 mg Tirzepatide vs Placebo; Midday Premeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -40.0, 95% CI 2-sided [-49.0 to -31.1]
Statistical Analysis 10: Comparison: 5 mg Tirzepatide vs Placebo; Midday 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -51.4, 95% CI 2-sided [-62.5 to -40.4]
Statistical Analysis 11: Comparison: 10 mg Tirzepatide vs Placebo; Midday 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -47.3, 95% CI 2-sided [-58.4 to -36.2]
Statistical Analysis 12: Comparison: 15 mg Tirzepatide vs Placebo; Midday 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -50.7, 95% CI 2-sided [-62.1 to -39.3]
Statistical Analysis 13: Comparison: 5 mg Tirzepatide vs Placebo; Evening Premeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -39.0, 95% CI 2-sided [-47.6 to -30.4]
Statistical Analysis 14: Comparison: 10 mg Tirzepatide vs Placebo; Evening Premeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -39.2, 95% CI 2-sided [-47.9 to -30.6]
Statistical Analysis 15: Comparison: 15 mg Tirzepatide vs Placebo; Evening Premeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -36.4, 95% CI 2-sided [-45.3 to -27.5]
Statistical Analysis 16: Comparison: 5 mg Tirzepatide vs Placebo; Evening 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -51.7, 95% CI 2-sided [-63.2 to -40.1]
Statistical Analysis 17: Comparison: 10 mg Tirzepatide vs Placebo; Evening 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -52.5, 95% CI 2-sided [-64.1 to -40.9]
Statistical Analysis 18: Comparison: 15 mg Tirzepatide vs Placebo; Evening 2-hour Postmeal; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -53.2, 95% CI 2-sided [-65.1 to -41.3]
Statistical Analysis 19: Comparison: 5 mg Tirzepatide vs Placebo; Bedtime; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -48.0, 95% CI 2-sided [-58.6 to -37.4]
Statistical Analysis 20: Comparison: 10 mg Tirzepatide vs Placebo; Bedtime; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -50.7, 95% CI 2-sided [-61.3 to -40.1]
Statistical Analysis 21: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -51.7, 95% CI 2-sided [-62.6 to -40.9]

7. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss ≥5%
Description: Percentage of Participants who Achieved Weight Loss ≥5%.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 121 | 118 | 116 | 112
Percentage of participants | 66.94 | 77.97 | 76.72 | 14.29
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.40, 95% CI 2-sided [6.43 to 23.94]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 21.13, 95% CI 2-sided [10.59 to 42.18]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 20.10, 95% CI 2-sided [10.09 to 40.04]

8. Secondary Outcome: Rate of Hypoglycemia With Blood Glucose <54 Milligram/Deciliter (mg/dL) [<3.0 Millimole/Liter (mmol/L)] or Severe Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with blood glucose <54mg/dL) (<3.0 mmol/L] or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. The rate of postbaseline hypoglycemia was estimated by negative binomial model: number of episodes = Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Prior Use of OAM (Yes, No) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline through end of safety follow-up (up to week 44)
Population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline value.
Measure: Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 121 | 119 | 120 | 115
Episodes/participant/365.25 days | 0.02 (0.002) | 0.02 (0.002) | 0.02 (0.002) | 0.04 (0.028)

9. Secondary Outcome: Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) of Tirzepatide
Description: Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) of Tirzepatide. AUC is a combined measure obtained from Week 7, 15 and 23, and a single averaged measure of AUC was reported.
Time Frame: Week 7, 15 and 23
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (h*ng/mL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 121 | 118 | 120
nanograms*hours per milliliter (h*ng/mL) | 86900 (25.4) | 171000 (26.2) | 252000 (23.3)

ADVERSE EVENTS:
Time Frame: Baseline to end of Safety follow-up (up to 44 weeks)
Description: All randomized participants who received at least one dose of study drug.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg of Tirzepatide as subcutaneous injection, once weekly.
- 10 mg Tirzepatide: Participants received 10 mg of Tirzepatide as subcutaneous injection, once weekly.
- 15 mg Tirzepatide: Participants received 15 mg of Tirzepatide as subcutaneous injection, once weekly.
- Placebo: Participants received placebo as subcutaneous injection, once weekly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121 | 0/121 | 1/115
Serious Adverse Events (participants affected / at risk) | 5/121 | 2/121 | 1/121 | 3/115
Other Adverse Events (participants affected / at risk) | 50/121 | 55/121 | 53/121 | 54/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=121) | 10 mg Tirzepatide (N=121) | 15 mg Tirzepatide (N=121) | Placebo (N=115)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=121) | 10 mg Tirzepatide (N=121) | 15 mg Tirzepatide (N=121) | Placebo (N=115)
Constipation (Gastrointestinal disorders) | 7 (11) | 6 (6) | 8 (9) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (21) | 17 (19) | 14 (20) | 9 (15)
Dyspepsia (Gastrointestinal disorders) | 11 (15) | 8 (12) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 14 (31) | 16 (82) | 22 (50) | 7 (8)
Vomiting (Gastrointestinal disorders) | 4 (6) | 3 (3) | 7 (9) | 2 (3)
Influenza (Infections and infestations) | 7 (7) | 3 (3) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (7) | 8 (13) | 8 (8) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 8 (9) | 10 (10) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (7) | 3 (3) | 31 (31)
Headache (Nervous system disorders) | 5 (9) | 4 (7) | 5 (8) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03954834/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03954834/SAP_001.pdf